CLINICAL TRIAL: NCT07070063
Title: Use of Virtual Reality in the Treatment of Various Types of Urinary Incontinence in Women
Brief Title: Virtual Reality for Urinary Incontinence in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Independent Public Health Care Center of the Ministry of the Interior and Administration in Wrocław (Unknown); Jan Dlugosz University in Czestochowa (Other); Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 49/2025
Record Dates: First submitted 2025-07-07; First posted 2025-07-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorder
Keywords: Virtual Reality; Rehabilitation; Pelvic Floor Muscle Training; Urinary incontinence; Women's health
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Group (Experimental): VR-Supported Pelvic Floor Training
  Interventions: Device: Virtual Reality Therapy; Device: Pelvic Floor Muscle Electrostimulation with EMG Biofeedback
- Control Group (Active Comparator): Conventional Pelvic Floor Training
  Interventions: Device: Pelvic Floor Muscle Electrostimulation with EMG Biofeedback

INTERVENTIONS:
Device: Virtual Reality Therapy — Eight sessions of virtual reality therapy will be administered over a two-week period (four sessions per week, each lasting 20 minutes). The intervention will be delivered using the VRTierOne device (Stolgraf®), which employs a head-mounted display to create a fully immersive environment. Through the integration of visual, auditory, and kinesthetic stimuli, the therapy provides a multi-sensory experience that can have calming and mood-enhancing effects, as well as support psychological engagement and motivation in the rehabilitation process. The virtual environment-designed as a therapeutic garden-is rich in symbols and metaphors derived from Ericksonian psychotherapy. The central element of this environment is the Garden of Revival, a metaphor for the patient's health. Once vibrant and full of life, the garden is now neglected and requires care and effort to be restored. Throughout the therapeutic process, the patient is guided by a symbolic narrative reflecting their individual
  Arms: VR Group
Device: Pelvic Floor Muscle Electrostimulation with EMG Biofeedback — Eight sessions of pelvic floor muscle electrostimulation combined with EMG biofeedback will be provided over a two-week period (four sessions per week). The intervention will be delivered using a specialized EMG-Biofeedback electrostimulation device equipped with a screen for real-time signal visualization. Vaginal electrodes will be used to ensure precise stimulation and accurate detection of pelvic floor muscle activity. During each 30-minute session, patients will receive symmetrical biphasic rectangular electrical impulses at a frequency of 50 Hz, with a 5-second stimulation phase followed by a 10-second rest period. The intensity of the stimulation will be individually adjusted to ensure both safety and comfort. The integrated biofeedback system will allow participants to observe their muscle activation patterns on the screen, enhancing their awareness and control of pelvic floor function and supporting the learning of correct activation during voluntary contractions.

SUMMARY:
This study evaluates the effectiveness of using virtual reality to support pelvic floor muscle training in women with urinary incontinence. The intervention aims to enhance patients' motivation, awareness, and exercise accuracy through real-time muscle visualization and immersive interaction. The project seeks to determine whether virtual reality-assisted therapy improves clinical outcomes compared to conventional approaches.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a common condition among women, negatively impacting quality of life, mental health, and social functioning. Although pelvic floor muscle training (PFMT) is an effective treatment, its success depends on proper technique and patient engagement-both of which are often insufficient due to limited education and challenges in exercise monitoring.

Virtual reality (VR) offers an innovative approach to support rehabilitation by providing real-time biofeedback, enhancing awareness of pelvic floor muscle function, and increasing motivation through immersive, interactive environments. Prior research suggests that VR can improve concentration, reduce therapy-related anxiety, and encourage active participation.

This study aims to evaluate the effectiveness of a VR-based system integrated with biofeedback in supporting PFMT for women with UI. Through real-time visualization of pelvic floor activity, the intervention may improve muscle control, exercise adherence, and clinical outcomes.

The project responds to the global trend of using digital tools in rehabilitation and addresses a gap in the literature concerning VR applications in urogynecology. While VR has shown promise in neurological and orthopedic rehabilitation, its potential in UI management remains underexplored. This trial seeks to generate evidence for its effectiveness and practical use in the treatment of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-80 years, who are at least 12 months post-menopausal,
* Diagnosed with urinary incontinence of grade I or IIa according to the ICS classification,
* No contraindications to participation (e.g., acute urinary tract infections, severe neurological disorders),
* Provision of written informed consent to participate in the research experiment.

Exclusion Criteria:

* Urinary incontinence of grade III or higher,
* Presence of significant neurological conditions affecting bladder control,
* Participation in other therapeutic interventions that could interfere with study outcomes,
* Pregnancy,
* Refusal or inability to provide informed consent.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Incontinence Quality of Life Questionnaire (I-QOL) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The I-QOL is a 22-item instrument designed to assess the impact of urinary incontinence on quality of life in women. It covers three domains: avoidance and limiting behaviors, psychosocial impacts, and social embarrassment. Items are rated on a 5-point Likert scale (1 = extremely to 5 = not at all). Scores are transformed into a scale ranging from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change from Baseline in the Incontinence Impact Questionnaire - Short Form (IIQ-7) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The IIQ-7 is a 7-item instrument that assesses the impact of urinary incontinence on various aspects of daily life, including physical activity, social relationships, emotional well-being, and travel. Each item is scored from 0 (not at all) to 3 (greatly), and total scores are standardized to a 0-100 scale. Higher scores indicate greater negative impact on quality of life.
Change from Baseline in the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, IUGA-Revised (PISQ-IR) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The PISQ-IR evaluates sexual function in women with urinary incontinence or pelvic organ prolapse. It includes separate domains for sexually active and inactive women, assessing aspects such as desire, satisfaction, and emotional impact. Higher scores in each domain indicate better sexual function and less impact of symptoms.
Change from Baseline in the Gaudenz Questionnaire for the Assessment of Urinary Incontinence Severity at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The Gaudenz Questionnaire assesses urinary incontinence severity through structured questions on leakage frequency, volume, triggers, and pad usage. It provides a detailed clinical profile of symptom severity, though not a single summary score.
Change from Baseline in the King's Health Questionnaire (KHQ) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The KHQ is a validated quality-of-life tool for individuals with urinary incontinence. It includes multiple domains such as general health perception, role limitations, physical limitations, social relationships, emotions, and sleep/energy. Each domain is scored on a 0-100 scale, with higher scores indicating greater impairment.
Change from Baseline in the Perceived Stress Questionnaire for Women (KPS) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The KPS is a validated Polish-language instrument designed to measure perceived stress in women. It evaluates subjective feelings of strain, tension, and inability to cope. Higher scores indicate higher levels of perceived stress.
Change from Baseline in Rosenberg Self-Esteem Scale (SES) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  The SES is a 10-item scale measuring global self-esteem. The Polish adaptation maintains the original structure and uses a 4-point Likert scale. Scores range from 10 to 40, with higher values reflecting higher self-esteem.
Change from Baseline in Presence and Grade of Pelvic Organ Prolapse (POP) at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  Pelvic organ prolapse (POP) will be evaluated using translabial ultrasound in the midsagittal plane. The presence and grade of anterior (cystocele), posterior (rectocele, enterocele), and apical (uterine or vaginal vault) prolapse will be determined relative to the inferoposterior margin of the symphysis pubis. POP grade will be classified according to the pelvic organ prolapse quantification system (POP-Q) or equivalent ordinal scale (Stage 0-IV). Higher stage values indicate more advanced prolapse severity.
Change from Baseline in Urethral Length and Structural Integrity at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  Urethral morphology will be assessed using transvaginal or translabial ultrasound. Structural integrity will be evaluated by identifying any abnormalities such as urethral diverticula, periurethral cysts, strictures, or focal discontinuities. Urethral length will be measured in millimeters (mm), from the bladder neck to the external urethral meatus. Structural defects will be reported categorically as present or absent. The presence of structural abnormalities is considered pathological. Shortened or disrupted urethral length may indicate structural compromise.
Change from Baseline in Bladder Wall Morphology at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  Bladder wall characteristics will be examined using transabdominal or translabial ultrasound. Thickness of the bladder wall will be measured in millimeters (mm) at the anterior wall with the bladder in a full state. Additional findings such as trabeculation, diverticula, or focal wall deformities will be documented as present or absent. Increased bladder wall thickness or the presence of structural abnormalities is considered indicative of chronic bladder dysfunction and is interpreted as adverse.
Change from Baseline in Bladder Neck Mobility at 2 weeks | From enrollment to the end of treatment at 2 weeks.
  Bladder neck mobility will be assessed using transvaginal or translabial ultrasound at rest and during the Valsalva maneuver. The degree of descent will be calculated as the displacement angle (in degrees) of the bladder neck relative to the pubic symphysis. An angle greater than 30-45° indicates hypermobility, which is considered pathological and commonly associated with stress urinary incontinence.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Kołodyńska, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland; Joanna Szczepańska-Gieracha, Professor, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland; Maciej Zalewski, PhD, Principal Investigator — Wroclaw Medical University (Poland); Waldemar Andrzejewski, Professor, Principal Investigator — Wroclaw University of Health and Sport Sciences, Poland
Locations (1):
- Independent Public Health Care Center of the Ministry of the Interior and Administration in Wrocław, Wroclaw, Lower Silesian Voivodeship, Poland